CLINICAL TRIAL: NCT02965248
Title: Multicenter, Randomized Controlled Trial Designed to Evaluate the Efficacy and Safety of Adjuvant Hyperthermic Intraperitoneal Chemotherapy (HIPEC) With Raltitrexed or Oxaliplatin Versus no HIPEC in Locally Advanced Colorectal Cancer (APEC Study)
Brief Title: Adjuvant Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Versus no HIPEC in Locally Advanced Colorectal Cancer (APEC Study)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guoxiang Cai, Associate Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1608163-15
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Locally Advanced Colorectal Cancer
Keywords: Locally advanced colorectal cancer; Hyperthermic intraperitoneal chemotherapy
MeSH Terms: interventions — Fluorouracil; Leucovorin; Capecitabine; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Active Comparator): Patients undergo radical resection of colorectal cancer (open/laparoscopic) and receive standard adjuvant systemic chemotherapy comprising mFOLFOX6/CapeOx/sLV5FU2/Cape. Systemic chemotherapy will continue for 6 months.
  Interventions: Drug: Standard adjuvant systemic chemotherapy
- Arm B (Experimental): Patients undergo radical resection of colorectal cancer (open/laparoscopic) and receive standard adjuvant systemic chemotherapy comprising mFOLFOX6/CapeOx/sLV5FU2/Cape. Systemic chemotherapy will continue for 6 months. Patients also undergo HIPEC with raltitrexed (3mg/m2) intraperitoneally for 60 minutes during surgery or within 10 days after the operation.
  Interventions: Drug: Standard adjuvant systemic chemotherapy; Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC) with raltitrexed
- Arm C (Experimental): Patients undergo radical resection of colorectal cancer (open/laparoscopic) and receive standard adjuvant systemic chemotherapy comprising mFOLFOX6/CapeOx/sLV5FU2/Cape. Systemic chemotherapy will continue for 6 months. Patients also undergo HIPEC comprising oxaliplatin (130mg/m2) intraperitoneally during surgery and hyperthermia for 30 minutes, following leucovorin calcium (20mg/m2 intravenously) and 5-FU (400 mg/m2 intravenously)
  Interventions: Drug: Standard adjuvant systemic chemotherapy; Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC) with oxaliplatin

INTERVENTIONS:
Drug: Standard adjuvant systemic chemotherapy — Patients undergo radical surgery with standard adjuvant systemic chemotherapy (mFOLFOX6/CapeOx/sLV5FU2/Cape).
  mFOLFOX6: oxaliplatin 85 mg/m2 IV d1 + leucovorin calcium 400 mg/m2 IV d1 + 5-FU 400 mg/m2 IV bolus d1 + 5-FU 2400 mg/m2 continuous IV over 46-48 hours d1-2. Repeat every two weeks for twelve cycles.
  CapeOx: oxaliplatin 130 mg/m2 IV d1 + capecitabine 1000mg/m2 po bid d1-14. Repeat every three weeks for eight cycles.
  sLV5FU2: leucovorin calcium 400 mg/m2 IV d1 + 5-FU 400 mg/m2 IV bolus d1 + 5-FU 2400 mg/m2 IV over 46-48 hours d1-2. Repeat every two weeks for twelve cycles.
  Cape: capecitabine 1000mg/m2 po bid d1-14. Repeat every three weeks for eight cycles.
  Other Names: adjuvant oxaliplatin, 5-FU, and leucovorin calcium (mFOLFOX6); adjuvant oxaliplatin and capecitabine (CapeOx); adjuvant 5-FU and leucovorin calcium (sLV5FU2); adjuvant capecitabine (Cape)
Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC) with raltitrexed — Raltitrexed (3 mg/m2) is added to the perfusate after attaining 42 degrees of inflow temperature and last for 60 minutes.
  Other Names: Intraperitoneal raltitrexed 3 mg/m2
  Arms: Arm B
Procedure: Hyperthermic intraperitoneal chemotherapy (HIPEC) with oxaliplatin — Before the beginning of HIPEC, 5-FU 400 mg/m2 and leucovorin calcium 20 mg/m2 will be administered intravenously to potentiate oxaliplatin activity. Oxaliplatin (130 mg/m2) is added to the perfusate after attaining 42 degrees inflow temperature with a total of 30 minutes perfusion time.
  Other Names: I.V. leucovorin calcium 20 mg/m2; I.V. 5-FU 400 mg/m2; Intraperitoneal oxaliplatin 130 mg/m2
  Arms: Arm C

SUMMARY:
This study is designed to evaluate the efficacy and safety of adjuvant hyperthermic intraperitoneal chemotherapy (HIPEC) with raltitrexed or oxaliplatin versus no HIPEC in locally advanced colorectal cancer

DETAILED DESCRIPTION:
Peritoneum is one of the common sites of metastasis in advanced stage colorectal cancer patients, resulting in a poor prognosis. Hyperthermic intraperitoneal chemotherapy (HIPEC) is effective to colorectal peritoneal metastasis and may play a significant role in reducing the risk of metachronous peritoneal metastasis among patients with locally advanced colorectal cancer. Oxaliplatin is routinely used for HIPEC in the Europe and Raltitrexed may be another ideal drug for HIPEC. The present phase II multicenter, randomized controlled trial is designed to evaluate the efficacy and safety of adjuvant HIPEC with raltitrexed or oxaliplatin versus no HIPEC in locally advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntarily and signed informed consent form
* Eastern Cooperative Oncology Group performance status of 0 to 1
* Life expectancy of more than 5 years
* Colorectal adenocarcinoma / mucinous adenocarcinoma / signet ring cell cancer confirmed by histopathology
* Stage T4NanyM0 cancer; or stage T3NanyM0 mucinous adenocarcinoma / signet ring cell cancer / adenocarcinoma with partly mucinous adenocarcinoma or signet ring cell cancer
* R0 resection of colorectal cancer
* Neutrophils (ANC) ≥ 1.5×10^9/L, Platelet count (Pt) ≥ 100× 10^9/L, Hemoglobin (Hb) ≥ 80 g/L, Hepatic function: ALT and AST ≤ 2.5 times upper limit of normal (ULN) and TBIL ≤ 1.5 times ULN, Renal function: creatinine ≤ 1.5 times ULN
* Use of an effective contraceptive for adults to prevent pregnancy

Exclusion Criteria:

* Rectal cancer below peritoneal reflection (≤ 8cm above the anal verge)
* Other malignant tumors within the past 5 years, except for skin basal cell carcinoma, or cervical carcinoma in situ, who survived from radical treatment
* Severe adhesion of peritoneal cavity impossible to separate
* Abdominal infection
* Allergic to raltitrexed, 5-FU, and oxaliplatin; Dihydropyrimidine dehydrogenase (DPD) enzyme deficiency
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior
* Drug addiction, Alcoholism or AIDS
* Impossible to tolerate the operation due to severe cardiac, lung, and vascular diseases
* Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
peritoneal metastasis rate | 3 years

SECONDARY OUTCOMES:
liver metastasis rate | 3 years
disease free survival | 3 years
overall survival | 5 years
quality of life questionnaire | 6 months
Toxicity by NCI CTCAE v.4.0 | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Guoxiang Cai, M.D. Ph.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China